CLINICAL TRIAL: NCT05707234
Title: Can we Avoid Intravenous Sedation in Patients Undergoing Knee Surgery Under Spinal Anesthesia? A Prospective Randomized Controlled Study Comparing Virtual Reality Hypnosis to Standard of Care
Brief Title: Virtual Reality Hypnosis in Total Knee Arthroplasty Under Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Michele Carella, Head of Clinic, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VRH.TKA
Record Dates: First submitted 2023-01-04; First posted 2023-01-31 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Arthroplasty Complications; Knee Osteoarthritis; Anesthesia Complication; Hypnotic; Anxiety Disorder; Sedation Complication
MeSH Terms: conditions — Osteoarthritis, Knee; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: prospective, single-center, randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): During the procedure, the patient in the control group receives pharmacological sedation, which is the standard of care currently practiced. Such sedation allows intraoperative anxiolysis, which is constantly required by patients in order to dissociate from their surroundings. Recall that total knee replacement surgery is extremely noisy, and the surrounding environment is itself an anxiety-provoking factor for the patient. Light to moderate, intraoperative sedation is carried out by intermittent boluses of midazolam 1 mg IV. Boluses are given every 5 minutes until a sedation level of -2 or -3 on the RASS (Richmond Agitation-Sedation Scale) scale is reached.
  Patients randomized to the control group will undergo perioperative anesthesia according to the current standards of care, without the addition of the VR headset or headphones.
  Interventions: Drug: Midazolam sedation
- VRH Group (Experimental): They will experience an underwater experience while listening to hypnotic script designed to induce a change in state of consciousness, increasing parasympathetic system tone and relaxation response, and reducing the perception of painful stimuli.
  During the whole procedure, an anesthesiologist will perform the usual cares, including closely monitoring, and will administrate intravenous sedation (midazolam) when necessary (see sedation protocol in the previous section).
  Interventions: Device: VRH; Drug: Midazolam sedation

INTERVENTIONS:
Device: VRH — The VR headset and headphones will be placed on patients after the spinal anesthesia, once the patient is positioned and the surgical drapes installed. Patients will then undergo a 120-minute Digital Sedation™ program (Aqua+© 120 Version 1.1 or subsequent version, Oncomfort SA, Waver, Belgium). They will experience an underwater experience while listening to hypnotic script designed to induce a change in state of consciousness, increasing parasympathetic system tone and relaxation response, and reducing the perception of painful stimuli. While the session is running, HCPs can see what is projected into the VRH headset on their Sedakit's X2 controller (i.e. the tablet connected to the glasses).
  Arms: VRH Group
Drug: Midazolam sedation — During the procedure, the patient in the control group receives pharmacological sedation, which is the standard of care currently practiced. Such sedation allows intraoperative anxiolysis, which is constantly required by patients in order to dissociate from their surroundings. Recall that total knee replacement surgery is extremely noisy, and the surrounding environment is itself an anxiety-provoking factor for the patient. Light to moderate, intraoperative sedation is carried out by intermittent boluses of midazolam 1 mg IV. Boluses are given every 5 minutes until a sedation level of -2 or -3 on the RASS (Richmond Agitation-Sedation Scale) scale is reached.

SUMMARY:
For many years, total knee arthroplasty (TKA) has been a common and effective procedure to treat chronic refractory joint pain. Although efforts must be pursued, as general anesthesia remains the main tendency for TKA. Currently, the standard of care to manage procedural anxiety is pharmacological sedation; i.e. the intravenous administration of additional anesthetic agents such as propofol or midazolam. However, pharmacological sedation has considerable undesirable side effects. Hence, risks of intraprocedural adverse events including respiratory depression, hemodynamic perturbations, or paradoxical effects such as hostility, aggression, and psychomotor agitation, are increased. The goal of this prospective, single-center, randomized controlled clinical trial is to systematically evaluate the impact of implementing a protocol of virtual reality hypnosis in patients undergoing total knee arthroplasty under spinal anesthesia.

DETAILED DESCRIPTION:
For many years, total knee arthroplasty (TKA) has been a common and effective procedure to treat chronic refractory joint pain. With a worldwide aging population, as well as a rising rate of obesity and related osteoarthritis, the utilization of TKA has considerably expanded over time, and this increase is expected to continue. Accordingly, healthcare systems are exploring various strategies to address this growing demand, while ensuring efficiency, cost-effectiveness and safety. Among these approaches, and based on several reports comparing the risks and benefits of general and regional anesthesia, a first attempt has been made to switch from performing TKAs under general to spinal anesthesia. Although efforts must be pursued, as general anesthesia remains the main tendency for TKA, results regarding spinal anesthesia are extremely encouraging. As such, spinal anesthesia has been associated with a decreased rate of complications, including wound infection, blood transfusions or mortality, and with reduced length of surgery and hospital stay.

Yet, while spinal anesthesia prevents procedural pain and ensures immobility of the operative territory, the patient is still awake, conscious of all the noises in the operating room, and can have a high level of intraoperative anxiety. Currently, the standard of care to manage procedural anxiety is pharmacological sedation; i.e. the intravenous administration of additional anesthetic agents such as propofol or midazolam. However, pharmacological sedation has considerable undesirable side effects. Hence, risks of intraprocedural adverse events including respiratory depression, hemodynamic perturbations, or paradoxical effects such as hostility, aggression, and psychomotor agitation, are increased. Moreover, it might lead to longer procedure duration or time to discharge, slower recovery, and postoperative delirium or cognitive dysfunction. In addition to these challenges, it becomes clear that procedural sedation directly impacts consumption of drugs such as opioids, triggering the highlighted risk of addiction.

In this context, new international guidelines for risk mitigation in pharmacological sedation have emerged. Both American and European anesthesia societies recommend particular caution in the use of sedative drugs, especially with benzodiazepines and in patients with obesity or obstructive sleep apnea, which are highly comorbid with knee osteoarthritis. However, only providing less, or even no sedatives at all, is not a valuable solution, as it would negatively impact patient comfort and satisfaction and negatively affect clinical workflow. Therefore, alternative, non-pharmacological interventions that would be able to reduce drug requirements and associated risks while ensuring a similar patient experience are being actively sought.

Among those approaches, there is currently a growing interest towards clinical hypnosis, a one-to-one delivered technique inducing "A state of consciousness involving focused attention and reduced peripheral awareness characterized by an enhanced capacity for response to suggestion". The hypnotic state involves the capacities of absorption (tendency to be fully involved in a mental experience), dissociation (a mental separation from the environment), and suggestibility (tendency to comply with hypnotic suggestions). When combined during surgery with conscious IV sedation and local or regional anesthesia, forming the so-called hypnosedation, clinical hypnosis is associated with improved perioperative safety and comfort as well as better clinical outcomes. More precisely, the use of clinical hypnosis during medical procedures has been shown to reduce pain, emotional distress and anxiety while preserving consciousness, spontaneous breathing, reflexes as well as hemodynamic and metabolic changes, to decrease the time spent in the operating room, and to have a beneficial impact on immediate recovery, characterized by reduced fatigue and postoperative nausea and vomiting (PONV). Furthermore, this technique allows to significantly reduce the administrated doses of IV sedation and the associated costs. Yet, several obstacles limit the use of hypnosedation as a standard of care in the operating/ procedure room: the need for continuous patient-side presence of trained professionals in the room (and the cost related to the mobilization of these professionals), the small number of cases per day one healthcare provider can handle, patient's language proficiency, as well as the heterogeneity of the responses to the hypnotic suggestions of patients themselves.

To overcome those limitations, Oncomfort has created Digital Sedation™ sessions, classified as Software as a Medical Device (SaMD), allowing to deliver clinical hypnosis - together with additional integrative therapeutic approaches - through virtual reality, a technique called Virtual Reality Hypnosis (VRH). Virtual reality (VR) is "a computer-generated simulation of a lifelike environment that can be interacted with in a seemingly real or physical way by a person, by means of responsive hardware such as a visor with screen or gloves with sensors. In the medical field, VR has been used as a non-pharmacological mean to alleviate pain, anxiety, and general discomfort during uncomfortable procedures. VR is thought to work by distracting patients from uncomfortable procedures: by giving the illusion of really going into the artificial world, VR is able to capture patient's attention away from the real environment. Accordingly, VR could strengthen the level of absorption and dissociation induced by clinical hypnosis, especially in low hypnotizable persons. Hence, VRH technology allows to deliver clinical hypnosis - and its related benefits- to a considerably greater number of patients. This automated way of delivering hypnosis responds to most of the limitations of the use of clinical hypnosis mentioned supra (e.g. availability of trained staff, language barrier,…).

To date, the Oncomfort's Digital Sedation™ is used in more than 100 hospitals, and more than 80 000 patients have already beneficiated from this type of VRH in daily clinical practice (e.g. interventional radiology, oncology, surgery,…). In line with its intended use, first studies have demonstrated that Digital Sedation™ reduces both experimental and clinical pain, as well as procedural anxiety. In addition, preliminary results indicate that it might replace midazolam during endoscopic urologic surgery, avoiding the respiratory side effects associated with pharmacological sedation. Over the last year, at the CHU of Liège, Digital Sedation™ has been offered to patients during orthopedic surgeries, demonstrating the feasibility of using VRH during TKAs performed under spinal anesthesia. While results seem to be positive in terms of performance of the procedure and patient satisfaction, the potential beneficial impact of this solution has not been systematically addressed yet. The goal of the present study is to objectify those effects, and in particular, to determine whether VRH can replace - at least in part- the intraoperative administration of midazolam, allowing to avoid its associated side effects while ensuring a similar patient's comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 yo and scheduled for elective knee arthroplasty under spinal anesthesia

Exclusion Criteria:

1. Low auditory and/or visual acuity that precludes the use of the device.
2. ASA status > 3
3. Head or face wounds precluding use of the device.
4. Schizophrenia or dissociative disorder.
5. Pregnancy.
6. Chronic renal insufficiency or severe hepatic insufficiency.
7. Non-proficiency in French (Research language).
8. Phobia of deep water.
9. Chronic pain and/or chronic analgesics consumption.
10. Medication affecting the autonomic nervous system.
11. Revision surgery.
12. Dizziness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Midazolam milligrams | 2 hours
  Sedation: Intravenous milligrams of midazolam administered during first 120 minutes of surgery to achieve a RASS (Richmond Agitation-Sedation Scale) of -2 or -3.

SECONDARY OUTCOMES:
Intensity of postoperative pain | 1 hour, 24 hours, 48 hours after surgery and one week later
  Pain (NRS 0-10)
Anxiety | 1 hour, 24 hours, 48 hours after surgery and one week later
  Anxiety (Numeric Rating Scale 0-10)
Anxiety | 1 hour, 24 hours, 48 hours after surgery and one week later
  Anxiety on State-Trait Anxiety Inventory scale (STAI-6)
Comfort | 1 hour, 24 hours, 48 hours after surgery and one week later
  Comfort during and after surgery (NRS 0-10)
Fatigue | 1 hour, 24 hours, 48 hours after surgery and one week later
  Fatigue (NRS 0-10)
Patient satisfaction | 5 minutes after surgery
  Patient satisfaction (global experience) Likert 1-5
Time perception | 5 minutes after surgery
  Patient's time perception (estimated duration of the surgery, i.e. duration between incision and suture)
Dissociation | 5 minutes after surgery
  Dissociation (NRS 0-10)
Anesthesiologist satisfaction | 5 minutes after surgery
  Anesthesiologist satisfaction (Likert 1-5)
Surgeon satisfaction | 5 minutes after surgery
  Surgeon satisfaction (Likert 1-5)
Nurse satisfaction | 5 minutes after surgery
  Nurse satisfaction (Likert 1-5)
QoR-15F | 1 hour, 24 hours, 48 hours after surgery and one week later
  Score on the quality of recovery, using the QoR-15F

OTHER OUTCOMES:
Length of Stay | 7 days after surgery
  Length of Stay (days)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carella M, Beck F, Quoilin C, Azongmo MM, Loheac A, Bonhomme VL, Vanhaudenhuyse A. Effect of virtual reality hypnosis on intraoperative sedation needs and functional recovery in knee arthroplasty: a prospective randomized clinical trial. Reg Anesth Pain Med. 2025 May 6;50(5):383-389. doi: 10.1136/rapm-2023-105261. PMID 38413184